CLINICAL TRIAL: NCT05539742
Title: Comparison of the Effect of Medium-Chain Fatty Acids and Long-Chain Fatty Acids on Postprandial Appetite and Lipemia
Brief Title: Comparison of the Effect of MCFA and LCFA on Postprandial Appetite and Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Shatha Hammad, Assistant Professor, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/6
Record Dates: First submitted 2022-06-13; First posted 2022-09-14 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Lipemia
Keywords: Postprandial lipemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Coconut Oil; Palm Oil

STUDY DESIGN:
Intervention Model Description: randomized crossover single-blinded intervention study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coconut oil (Active Comparator): The coconut oil will be given to each participant in the amount of 40 g, which will be incorporated into biscuits. Each participant will have ten minutes to consume biscuits with 250 ml of water. No other food will be consumed during the study period (6 hours). After that, participants will be allowed an ad libitum intake of standard meals. Each meal will be weighed before and after it is consumed, with the amount of food ingested being calculated. Then the participants will take the other treatment after a 1-week washout interval.
  Interventions: Dietary Supplement: Coconut oil
- Palm oil (Active Comparator): The palm oil will be given to each participant in the amount of 40 g, which will be incorporated into biscuits. Each participant will have ten minutes to consume biscuits with 250 ml of water. No other food will be consumed during the study period (6 hours). After that, participants will be allowed an ad libitum intake of standard meals. Each meal will be weighed before and after it is consumed, with the amount of food ingested being calculated. Then the participants will take the other treatment after a 1-week washout interval.
  Interventions: Dietary Supplement: Palm oil

INTERVENTIONS:
Dietary Supplement: Coconut oil — Coconut oil will be given to each participant in the amount of 40 g, which will be incorporated into biscuits.
  Arms: Coconut oil
Dietary Supplement: Palm oil — Palm oil will be given to each participant in the amount of 40 g, which will be incorporated into biscuits.
  Arms: Palm oil

SUMMARY:
The main objective is to investigate if foods high in coconut oil (MCFA) or palm oil (LCFA) have different impacts on postprandial blood lipid levels and appetite via a visual analog scale (VAS).

DETAILED DESCRIPTION:
Postprandial lipemia has been recognized as a cardiovascular disease risk factor. The rate of postprandial triglyceride production and clearance in the blood, as well as the appetite, are influenced by the quality of the food consumed, such as the length of saturated fatty acids. The study will include 24 healthy adults ranging in age from 18 to 40 years old, of both sexes and it will be conducted at the University of Jordan. The study will involve two experimental test days, each separated by at least a week of washout interval, and each test day will last for 6 hours. All subjects will be randomly assigned to one of the experimental meals using computer-generated tables. Blood serum samples (2 mL) will be taken after an overnight fast and 2, 4, and 6 hours after eating the meals, and blood lipid profiles [total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglyceride (TG)] will be examined in a private lab. After that, participants will be allowed an ad libitum intake of standard meals. Each meal will be weighed before and after it is consumed, with the amount of food ingested being calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years
* Males and females
* Apparently healthy
* Fasting triglyceride (TG) < 2.5 mmol/L or 222 mg/dl at the time of screening.
* Body mass index (BMI) in normal range (18.5-24.9).
* Stable weight for at least 3 months

Exclusion Criteria:

* Consumption of lipid-lowering drugs or any medication that might affect appetite.
* Consumption of any supplement that may affect lipid metabolism or appetite on a regular basis for the past month.
* Regular consumption of two or more fish meals a week over the previous month.
* A history of diabetes, gastrointestinal , liver disease, congestive heart failure, stroke, myocardial infarction, coronary artery bypass graft or established atherosclerotic disease.
* Current smokers
* Pregnant , breastfeeding, postmenopausal or suffer from polycystic ovary syndrome (PCOS)
* Athlete
* Being on a diet or lifestyle changes for the past month.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements ( Height) | baseline, pre-intervention, 1 day for each participant /during 3 months
  Standing height, without footwear, will be taken using stadiometer to the nearest 5mm
Anthropometric measurements (Weight) | baseline, pre-intervention, 1 day for each participant /during 3 months
  Bioelectrical impedance will be used to determine body weight
Anthropometric measurements (waist circumference) | baseline, pre-intervention, 1 day for each participant /during 3 months
  Waist circumference (WC) will be measured at the midway between the lowest ribs and the iliac crest using a standard tape to the nearest 1 cm
Anthropometric measurements (percentage body fat) | baseline, pre-intervention,1 day for each participant /during 3 months
  Bioelectrical impedance will be used to determine body composition
Biochemical measurements (Total cholesterol (TC)) | After the intervention / up to 3 months from collecting the samples
  Up to 6 hours
Biochemical measurements (Low density lipoprotein cholesterol (LDL)) | Up to 6 hours
  Low-density lipoprotein cholesterol test will be performed after an overnight fast and 2, 4, and 6 hours after eating the meals
Biochemical measurements ( High density lipoprotein cholesterol (HDL)) | Up to 6 hours
  High-density lipoprotein cholesterol test will be performed after an overnight fast and 2, 4, and 6 hours after eating the meals
Biochemical measurements (Triglyceride (TG)) | Up to 6 hours
  Triglyceride test will be performed after an overnight fast and 2, 4, and 6 hours after eating the meals
Dietary intake (3-days food record) | one day
  Participants will be asked to fill out a food record to track changes in their (intake) appetite

CONTACTS AND LOCATIONS:
Overall Officials: Shatha S Hammad, PhD, Principal Investigator — The University of Jordan
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin G, Ferguson JJ, Thota RN, Singh H, Burrows T, Garg ML. Postprandial lipaemia following consumption of a meal enriched with medium chain saturated and/or long chain omega-3 polyunsaturated fatty acids. A randomised cross-over study. Clin Nutr. 2021 Feb;40(2):420-427. doi: 10.1016/j.clnu.2020.06.027. Epub 2020 Jul 1. PMID 32684486
- [Background] Abedi E, Sahari MA. Long-chain polyunsaturated fatty acid sources and evaluation of their nutritional and functional properties. Food Sci Nutr. 2014 Sep;2(5):443-63. doi: 10.1002/fsn3.121. Epub 2014 Jun 29. PMID 25473503
- [Background] Behrouz V, Yari Z. A review on differential effects of dietary fatty acids on weight, appetite and energy expenditure. Crit Rev Food Sci Nutr. 2022;62(8):2235-2249. doi: 10.1080/10408398.2020.1852172. Epub 2020 Dec 1. PMID 33261509
- [Background] Boateng L, Ansong R, Owusu WB, Steiner-Asiedu M. Coconut oil and palm oil's role in nutrition, health and national development: A review. Ghana Med J. 2016 Sep;50(3):189-196. PMID 27752194
- [Background] Bozzetto L, Della Pepa G, Vetrani C, Rivellese AA. Dietary Impact on Postprandial Lipemia. Front Endocrinol (Lausanne). 2020 Jul 7;11:337. doi: 10.3389/fendo.2020.00337. eCollection 2020. PMID 32733374
- [Background] Dias CB, Moughan PJ, Wood LG, Singh H, Garg ML. Postprandial lipemia: factoring in lipemic response for ranking foods for their healthiness. Lipids Health Dis. 2017 Sep 18;16(1):178. doi: 10.1186/s12944-017-0568-5. PMID 28923057
- [Background] Folwaczny A, Waldmann E, Altenhofer J, Henze K, Parhofer KG. Postprandial Lipid Metabolism in Normolipidemic Subjects and Patients with Mild to Moderate Hypertriglyceridemia: Effects of Test Meals Containing Saturated Fatty Acids, Mono-Unsaturated Fatty Acids, or Medium-Chain Fatty Acids. Nutrients. 2021 May 20;13(5):1737. doi: 10.3390/nu13051737. PMID 34065380
- [Background] Karupaiah T, Tan CH, Chinna K, Sundram K. The chain length of dietary saturated fatty acids affects human postprandial lipemia. J Am Coll Nutr. 2011 Dec;30(6):511-21. doi: 10.1080/07315724.2011.10719997. PMID 22331686
- [Background] Kaviani S, Cooper JA. Appetite responses to high-fat meals or diets of varying fatty acid composition: a comprehensive review. Eur J Clin Nutr. 2017 Oct;71(10):1154-1165. doi: 10.1038/ejcn.2016.250. Epub 2017 Jan 18. PMID 28098139
- [Background] Khaw KT, Sharp SJ, Finikarides L, Afzal I, Lentjes M, Luben R, Forouhi NG. Randomised trial of coconut oil, olive oil or butter on blood lipids and other cardiovascular risk factors in healthy men and women. BMJ Open. 2018 Mar 6;8(3):e020167. doi: 10.1136/bmjopen-2017-020167. PMID 29511019
- [Background] Maher T, Sampson A, Goslawska M, Pangua-Irigaray C, Shafat A, Clegg ME. Food Intake and Satiety Response after Medium-Chain Triglycerides Ingested as Solid or Liquid. Nutrients. 2019 Jul 17;11(7):1638. doi: 10.3390/nu11071638. PMID 31319633
- [Background] Ma WY, Yang CY, Shih SR, Hsieh HJ, Hung CS, Chiu FC, Lin MS, Liu PH, Hua CH, Hsein YC, Chuang LM, Lin JW, Wei JN, Li HY. Measurement of Waist Circumference: midabdominal or iliac crest? Diabetes Care. 2013 Jun;36(6):1660-6. doi: 10.2337/dc12-1452. Epub 2012 Dec 28. PMID 23275359
- [Background] Moneeb AHM, Hammam ARA, Ahmed AKA, Ahmed ME, Alsaleem KA. Effect of fat extraction methods on the fatty acids composition of bovine milk using gas chromatography. Food Sci Nutr. 2021 May 4;9(6):2936-2942. doi: 10.1002/fsn3.2252. eCollection 2021 Jun. PMID 34136161
- [Background] Montoya C, Cochard B, Flori A, Cros D, Lopes R, Cuellar T, Espeout S, Syaputra I, Villeneuve P, Pina M, Ritter E, Leroy T, Billotte N. Genetic architecture of palm oil fatty acid composition in cultivated oil palm (Elaeis guineensis Jacq.) compared to its wild relative E. oleifera (H.B.K) Cortes. PLoS One. 2014 May 9;9(5):e95412. doi: 10.1371/journal.pone.0095412. eCollection 2014. PMID 24816555
- [Background] Panth N, Abbott KA, Dias CB, Wynne K, Garg ML. Differential effects of medium- and long-chain saturated fatty acids on blood lipid profile: a systematic review and meta-analysis. Am J Clin Nutr. 2018 Oct 1;108(4):675-687. doi: 10.1093/ajcn/nqy167. PMID 30239550
- [Background] Panth N, Dias CB, Wynne K, Singh H, Garg ML. Medium-chain fatty acids lower postprandial lipemia: A randomized crossover trial. Clin Nutr. 2020 Jan;39(1):90-96. doi: 10.1016/j.clnu.2019.02.008. Epub 2019 Feb 16. PMID 30824268
- [Background] Pirillo A, Norata GD, Catapano AL. Postprandial lipemia as a cardiometabolic risk factor. Curr Med Res Opin. 2014 Aug;30(8):1489-503. doi: 10.1185/03007995.2014.909394. Epub 2014 May 2. PMID 24673475
- [Background] Schonfeld P, Wojtczak L. Short- and medium-chain fatty acids in energy metabolism: the cellular perspective. J Lipid Res. 2016 Jun;57(6):943-54. doi: 10.1194/jlr.R067629. Epub 2016 Apr 14. PMID 27080715
- [Background] Tan J, McKenzie C, Potamitis M, Thorburn AN, Mackay CR, Macia L. The role of short-chain fatty acids in health and disease. Adv Immunol. 2014;121:91-119. doi: 10.1016/B978-0-12-800100-4.00003-9. PMID 24388214
- [Background] Teng KT, Chang CY, Kanthimathi MS, Tan AT, Nesaretnam K. Effects of amount and type of dietary fats on postprandial lipemia and thrombogenic markers in individuals with metabolic syndrome. Atherosclerosis. 2015 Sep;242(1):281-7. doi: 10.1016/j.atherosclerosis.2015.07.003. Epub 2015 Jul 7. PMID 26232169
- [Background] Tvrzicka E, Kremmyda LS, Stankova B, Zak A. Fatty acids as biocompounds: their role in human metabolism, health and disease--a review. Part 1: classification, dietary sources and biological functions. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2011 Jun;155(2):117-30. doi: 10.5507/bp.2011.038. PMID 21804620
- [Background] Zentek J, Buchheit-Renko S, Ferrara F, Vahjen W, Van Kessel AG, Pieper R. Nutritional and physiological role of medium-chain triglycerides and medium-chain fatty acids in piglets. Anim Health Res Rev. 2011 Jun;12(1):83-93. doi: 10.1017/S1466252311000089. PMID 21676342
- [Derived] Jadallah R, Hammad SS. Comparison of the effect of medium-chain fatty acids and long-chain fatty acids on postprandial appetite and lipemia: a randomised crossover trial. BMJ Nutr Prev Health. 2024 Dec 11;7(2):e001029. doi: 10.1136/bmjnph-2024-001029. eCollection 2024. PMID 39882282